CLINICAL TRIAL: NCT02984124
Title: Communication During Hospitalization About Resuscitation Trial
Acronym: CHART
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: University of Washington (Other); Medical University of South Carolina (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Renee Stapleton, Associate Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHRMS 16-227
Record Dates: First submitted 2016-11-28; First posted 2016-12-06 (Estimated); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Severe Life-limiting COPD; Severe Life-limiting Heart Failure; Severe Life-limiting Cirrhosis; Severe Life-limiting Malignancy; Severe Functional Impairment; End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Participants (n= approximately 100 plus family members) who are randomized to the intervention arm of the study will participate in a discussion about CPR with a study doctor.
  Interventions: Behavioral: Informed Assent Discussion
- Usual Care with Attention Control (Placebo Comparator): Participants (n= approximately 100 plus family members) who are randomized to the usual care arm will receive a friendly visit in the hospital from research personnel to ask if they have any questions or concerns. Follow up assessments and time windows will be explained. Importance of their participation in the study will be emphasized.
  Interventions: Behavioral: Usual Care with Attention Control

INTERVENTIONS:
Behavioral: Informed Assent Discussion — Participants randomized to the intervention arm will participate in a discussion about CPR with a study doctor that follows these steps:
  1. Patient's values and preferences for therapies and outcomes elicited from patient and family; overall therapeutic goals formulated
  2. Description of CPR and dying process provided
  3. Personalized explanation provided about probable lack of achieving any reasonable therapeutic goal with CPR (i.e. why s/he is a poor candidate for CPR due to underlying illness)
  4. Patient and family informed that due to severe underlying illness and high likelihood that CPR will be burdensome/harmful and will not provide benefit, CPR will not be offered unless they disagree (except in rare circumstance where overall therapeutic goals from step 1 are to preserve life regardless of quality of that life) Assessment of patient's and family's understanding of issues discussed; patients may actively disagree and request CPR be performed, but CPR not explicitly offered
  Arms: Intervention
Behavioral: Usual Care with Attention Control — Participants who are randomized to the usual care arm will receive a friendly visit in the hospital from research personnel to ask if they have any questions or concerns. Follow up assessments and time windows will be explained. Importance of their participation in the study will be emphasized.
  Arms: Usual Care with Attention Control

SUMMARY:
This multicenter RCT of 200 hospitalized patients and their family members evaluates an "informed assent" approach to discussing cardiopulmonary resuscitation, compared to usual care, in older seriously ill hospitalized patients with severe life-limiting illness or severe functional impairment.

DETAILED DESCRIPTION:
Increasing evidence suggests that high quality palliative care in older patients improves quality of care, patient and family satisfaction, and costs of care. However, while some specific palliative care interventions have been investigated, exactly how we should provide this care remains unclear. One important component of high quality provider-patient communication is discussing cardiopulmonary resuscitation (CPR) within the context of the patient's values and goals of care. Unfortunately, these conversations are often rushed, focused only on the procedure rather than the patient's goals and values, and CPR is often offered as if a choice on a menu. Elderly hospitalized patients are unlikely to have made decisions about CPR prior to hospitalization, and these discussions often leave patients and families feeling burdened, stressed, and concerned. Outcomes after in-hospital CPR in chronically ill older patients continue to be very poor, despite decades of efforts toward improvement.

The investigators aim to change the paradigm of CPR discussions with older adults unlikely to benefit from CPR. This study is a randomized controlled trial comparing an innovative "informed assent" approach to discussing CPR versus usual care with attention control for older hospitalized adults with life-limiting illness or severe functional impairment, enrolling patients and family members at three different study sites. Informed assent includes: 1) eliciting values and goals, 2) explaining CPR in the context of illness, and 3) a caring statement that the patient should not receive CPR if values include avoiding burdensome therapies unlikely to provide benefit. Thus, the provider can elicit values, convey information, and state an assessment, while allowing the patient or family to disagree. The investigators hypothesize that informed assent will improve quality of and satisfaction with communication about CPR; reduce the burden of potentially harmful CPR discussions, including reduced patient and family symptoms of depression and anxiety; and reduce intensity of care and health care utilization. The intervention builds on prior work investigating CPR outcomes in older adults and performing pilot studies of the informed assent intervention in both inpatients and outpatients.

ELIGIBILITY:
Inclusion Criteria:

1. >65 years old
2. English speaking
3. Must have one or more of the following:

   1. Chronic life-limiting illness with median survival <2 years defined as: 1) metastatic cancer or inoperable lung cancer; 2) COPD requiring oxygen; 3) New York Heart Association Class III or IV heart failure, 4) Child's Class C cirrhosis or MELD score of >20, 5) End-stage renal disease (must be on dialysis and ≥ 75 years old), 6) Advanced pulmonary fibrosis/interstitial lung disease, 7) Advanced pulmonary hypertension
   2. Severe functional impairment defined as dependence with >4 activities of daily living (ADLs) on Katz Index of Independence in ADLs.

Exclusion Criteria:

1. Has already definitively chosen DNR status
2. Unable to provide informed consent
3. Refused consent
4. Currently listed on a transplant list (awaiting transplant)
5. Inappropriate for study enrollment per clinician
6. Known to have a left ventricular assist device (LVAD)
7. Research team unavailable
8. Patient discharged from hospital prior to enrollment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 182 (Actual)
Dates: Start 2016-12; Primary Completion 2023-03 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Communication Questionnaire (QOCQ), slightly modified to focus on communication about cardiopulmonary resuscitation | Study day 5 +/- 1 or hospital discharge, whichever is earlier
  Patient-Assessed Quality of Communication about CPR

SECONDARY OUTCOMES:
Quality of Communication Questionnaire (QOCQ), slightly modified to focus on communication about cardiopulmonary resuscitation | Study day 5 +/- 1 or hospital discharge, whichever is earlier
  Family-Assessed Quality of Communication about CPR
5-question communication domain of the CANHELP Questionnaire, slightly modified to focus on communication about cardiopulmonary resuscitation | Study day 5 +/- 1 or hospital discharge, whichever is earlier
  Patient-Assessed Satisfaction with Communication about CPR
5-question communication domain of the CANHELP Questionnaire, slightly modified to focus on communication about cardiopulmonary resuscitation | Study day 5 +/- 1 or hospital discharge, whichever is earlier
  Family-Assessed Satisfaction with Communication about CPR
Hospital Anxiety and Depression Survey (HADS) | Study day 5 +/- 1 or hospital discharge (whichever is earlier), 3 months, and 6 months
  Patient Depressive and Anxiety Symptoms
Hospital Anxiety and Depression Survey (HADS) | Study day 5 +/- 1 or hospital discharge (whichever is earlier), 3 months, and 6 months
  Family Depressive and Anxiety Symptoms
Do-Not-Resuscitate Orders (yes/no) | Study day 5 +/- 1 or hospital discharge (whichever is earlier), 3 months, and 6 months
Time to Do-Not-Resuscitate Orders | To 6 months post-randomization
Admission to the intensive care unit (ICU) 9yes/no) | Measured at the time hospital discharge, which will likely occur at an average of 6 days after admission, but will be assessed for up to 6 months.
ICU length of stay (days) | Measured at the time hospital discharge, which will likely occur at an average of 6 days after admission, but will be assessed for up to 6 months.
Tracheostomy placement (yes/no) | Measured at the time hospital discharge, which will likely occur at an average of 6 days after admission, but will be assessed for up to 6 months.
Gastrostomy tube placement (yes/no) | Measured at the time hospital discharge, which will likely occur at an average of 6 days after admission, but will be assessed for up to 6 months.
Receipt of mechanical ventilation (yes/no) | Measured at the time hospital discharge, which will likely occur at an average of 6 days after admission, but will be assessed for up to 6 months.
Receipt of renal replacement therapy (yes/no) | Measured at the time hospital discharge, which will likely occur at an average of 6 days after admission, but will be assessed for up to 6 months.
Receipt of cardiopulmonary resuscitation (yes/no) | Measured at the time hospital discharge, which will likely occur at an average of 6 days after admission, but will be assessed for up to 6 months.
Cost of health care after initial hospitalization | 3 months and 6 months post-randomization
  Repeat hospital admissions, ICU admissions, nursing home says, hospice care stays, and use of home health care will be assessed, and if they occurred, duration will be recorded. A standardized value (costs, not charges) will be applied to these measures to determine overall cost.
Mortality (dead or alive) | To 6 months post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Renee Stapleton, MD PhD, Principal Investigator — University of Vermont
Locations (4):
- United States (4):
  - University of North Carolina, Chapel Hill, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Vermont, Burlington, Vermont
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
This study includes quantitative data that the investigators plan to share with other researchers with interests in the quality of care provided to older hospitalized seriously ill patients and their families. De-identified questionnaire data, medical record data, and administrative data will be made available in the form of datasets with no personally identifying characteristics retained, to protect the identity of the respondents.